CLINICAL TRIAL: NCT00254774
Title: Pilot Study of the Efficacy and Safety of Quetiapine Compared With Valproate in the Treatment of Patients With Bipolar Disorder and Rapid Cycling: an Open Trial
Brief Title: Efficacy and Safety of Quetiapine Compared With Valproate in the Treatment of Patients With Bipolar Disorder and Rapid Cycling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5077/9061; D1441C09061
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2007-12-18 (Estimated); Status verified 2007-12

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder I or II with Rapid Cycling
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Valproic Acid

INTERVENTIONS:
Drug: quetiapine fumarate or valproate

SUMMARY:
The purpose of the study is to evaluate the efficacy of quetiapine compared to valproate during a 12 month treatment period in subjects with Bipolar Disorder I or II with Rapid Cycling.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, men and women aged ³18 to £65 years with diagnosis of DSM-IV criteria for bipolar I or II disorder, most recent episode manic, hypomanic, mixed or depressive with Rapid Cycling.

Exclusion Criteria:

* Substance or alcohol dependence, female patients who are pregnant, lactating or at risk of pregnancy, diagnosis of schizophrenia or borderline personality disorder or antisocial personality disorder, history of seizure disorder, acute suicidal or external aggressive behaviour, legal incapacity or indication for treatment against the will of the patient by law.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-01; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Number of clinically relevant recurrences of depression or mania. Recurrence is defined by a change in LCM-C/P to moderate or severe or by 2 or more steps. End of an episode is defined as reduction to mild or baseline or by 2 or more steps.

SECONDARY OUTCOMES:
Absolute change from baseline on the (recalculated) HAM-D, YMRS, MADRS, total score. Absolute change from baseline on the CGI-BP severity score per dimension (mania, depression, overall bipolar illness).

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Germany Medical Director, MD, Study Director — AstraZeneca
Locations (3):
- Germany (3):
  - Research Site, Berlin
  - Research Site, Freiburg im Breisgau
  - Research Site, München